CLINICAL TRIAL: NCT03704480
Title: Durvalumab Plus Tremelimumab Combination Immunotherapy With or Without Weekly Paclitaxel in Patients With Advanced Biliary Tract Carcinoma (BTC) After Failure of Platinum-based Chemotherapy: a Randomized Non-comparative Two-arm Phase II Study
Brief Title: Durvalumab + Tremelimumab ± Paclitaxel in Advanced BTC After Platinum Chemotherapy.
Acronym: IMMUNO-BIL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMMUNO-BIL D18-1 PRODIGE 57
Record Dates: First submitted 2018-09-28; First posted 2018-10-12 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Advanced Biliary Tract Carcinoma
Keywords: Immunotherapy
MeSH Terms: interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amended ARM A (Experimental): One cycle equals 4 weeks (D1=D28);
  Durvalumab: 1,500 mg by IV infusion on D1, until progression or unacceptable toxicity or withdrawal of consent.
  Tremelimumab: 300 mg by IV infusion on D1 at cycle 1 only.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: Durvalumab — 1500mg by intravenous (IV) infusion on D1 until progression or unacceptable toxicity or withdrawal of consent
  Other Names: MEDI4736
Drug: Tremelimumab — 300mg by IV infusion on D1 at cycle 1 only
  Other Names: CP-675

SUMMARY:
IMMUNO-BIL is a non-comparative randomized 1:1 phase II study. This study will assess the efficacy and safety of the combination of durvalumab plus tremelimumab with or without weekly paclitaxel in patients with advanced BTC after failure of platinum-based chemotherapy.

On the 25th June 2019, the maximum DLT event number was reached (6/10) in the durvalumab plus tremelimumab combination with paclitaxel Arm (Arm B). According to the Pocock boundary described in the protocol, GERCOR has updated the study to discontinue enrollment in Arm B (durvalumab plus tremelimumab with paclitaxel) . No safety concerns were raised by the IDMC in Arm A. Consequently, the study will resume with Arm A (durvalumab plus tremelimumab) only, without randomization.

Discontinuation of ARM B(June 2019): Durvalumab plus tremelimumab plus paclitaxel

One cycle equals 4 weeks (D1=D28); Durvalumab: 1,500 mg by IV infusion on D1, until progression or unacceptable toxicity or withdrawal of consent.

Tremelimumab: 75 mg by IV infusion on D1 for the first 4 cycles. Paclitaxel: 80 mg/m2, every week for 3 weeks (D1-D8-D15), by IV infusion, until progression or unacceptable toxicity or withdrawal of consent (at least 6 cycles, at the discretion of the investigator).

December 2020: Tremelimumab dosage modification based on the results of the Study 22 study (Kelley RK, et al. ASCO20 Virtual Scientific Program 2020) showing increased efficacy (response rate and progression-free survival) without safety concerns with one dose of tremelimumab 300 mg (cycle 1) instead of four doses of 75 mg (cycle 1 to cycle 4) in combination with durvalumab 1,500 mg Q4W in hepatocellular carcinoma. Following these results, we have changed the tremelimumab 75 mg x 4 schedule for the 300 mg x 1 schedule. The inclusion of 106 additional patients will be required to adequately evaluate the efficacy of this administration schedule.

ARM A : Durvalumab plus tremelimumab ( patients included before 31/12/2020) One cycle equals 4 weeks (D1=D28);

Durvalumab: 1,500 mg by IV infusion on D1, until progression or unacceptable toxicity or withdrawal of consent.

Tremelimumab: 75 mg by IV infusion on D1 for the first 4 cycles.

DETAILED DESCRIPTION:
Biliary tract carcinoma (BTC, adenocarcinoma in more than 90% of cases) is the second primary liver tumor in incidence after hepatocellular carcinoma (2,000 new cases/year in France).

The prognosis of biliary malignancies is poor, with a 5-year overall survival rate (OS) of about 10-15%, most often due to late diagnosis, at an advanced stage.

In advanced BTC, the gemcitabine plus platinum (cisplatin [GEMCIS] or oxaliplatin [GEMOX]) doublet of chemotherapy is the standard first-line treatment and no targeted therapy has been validated in this indication to date. There is no second-line therapeutic standard; chemotherapy (mainly, 5-FU-based combination) yields limited median progression-free survival (PFS) and OS of abouty 2-3 months and 6-7 months respectively, justifying the exploration of new therapeutic options.

Immune therapies (mainly, immune checkpoint inhibitors [ICI]) have opened new opportunities in cancer therapy. Hence, anti-CTLA-4 and anti-PD-1/PD-L1 monoclonal antibodies (mAb) have demonstrated robust clinical activity and obtained FDA approval in several cancers. Recent data showed encouraging results with anti-PD-1 mAb as a monotherapy in PD-L1-positive pre-treated advanced BTC. The effects of ICI in combination with second-line chemotherapy in patients with advanced BTC have not been explored to date.

Platinum salts can induce "immunogenic cell death". Therefore, previous treatment with platinum may increase tumor immunogenicity and sensitivity to immune therapy, particularly, ICI. The second-line setting after failure of platinum-based chemotherapy may then be an optimal biological context for testing immune therapy in advanced BTC.

Durvalumab is a human immunoglobulin (Ig) G1 kappa (IgG1κ) anti-PD-L1 mAb. Tremelimumab is a human IgG2 anti-CTLA-4 mAb. Paclitaxel is a chemotherapy belonging to the taxane family. Taxanes may enhance the effect of immunotherapy by increasing the sensitivity of the tumor and activating the immune system. Taxanes are used in some patients with advanced biliary cancer.

These data suggest that BTC may be a good candidate for immune therapy. The combination of anti-CTL4 and anti-PD1/PD-L1 mAb is expected to be active in both immune-inflamed and non-inflamed BTC, and in PD-L1 high and low tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the patient prior to performing any protocol-related procedures, including screening evaluations.
2. Willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
3. Histologically or cytologically proven BTC (extrahepatic CCA, intrahepatic CCA, or gallbladder carcinoma).
4. Failure (documented progression or toxicity) of previous platinum-based (cisplatin or oxaliplatin) therapy (e.g. GEMCIS, GEMOX, FOLFIRINOX) Note: a maximum of 1 previous chemotherapy line is allowed; maintenance therapy with chemotherapy or targeted agent, except immunotherapy, will be permitted.
5. Age ≥ 18 years at the time of study entry.
6. ECOG PS 0-1.
7. Recurrent or advanced disease not amenable to surgery, radiation, or combined modality therapy with curative intent (previous resection of primary tumor allowed).
8. Measurable or evaluable (radiologically detectable disease which does not fulfill RECIST criteria for measurable disease) lesions according to RECIST v1.1 criteria (CT-scan < 3 weeks).
9. Have tissue from an archival tissue sample that has been identified and confirmed as available for study, or newly obtained core or excisional biopsy of a tumor lesion.
10. Adequate organ function, as defined by the following:

    * Serum aspartate aminotransferase (AST) and serum alanine aminotransferase (ALT) < 3 x upper limit of normal (ULN)
    * Total serum bilirubin < 1.5 ULN
    * Prothrombin ratio > 70%
    * Serum albumin ≥ 28 g/L
    * Hemoglobin ≥ 9.0 g/dl
    * White blood cell count (WBC) ≥ 3,000/μL
    * Absolute neutrophil count (ANC) ≥ 1,500/μL
    * Platelets ≥ 100,000/μL
    * Serum creatinine ≤ 1.5 ULN or creatinine clearance > 50 mL/min (MDRD).
11. Body weight > 40 kg.
12. Any other prior therapy directed at the malignant tumor, including chemotherapy, chemoembolization therapy, molecular targeted therapy (including antiangiogenics), and radiotherapy, must be discontinued at least 2 weeks prior to registration and at least 3 weeks before day 1 on trial.
13. Life expectancy ≥ 3 months.
14. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).

    Women ≥ 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

    Women participants of childbearing potential must have a negative serum pregnancy test within the 7 days prior to the first treatment administration. Both women participants of childbearing potential and men participants who are sexually active with women of childbearing potential must agree to use a reliable method of birth control (i.e. pregnancy rate < 1% per year); women of childbearing potential will be instructed to adhere to contraception for a period of 180 days after the last dose of durvalumab and tremelimumab or 90 days after the last dose of durvalumab monotherapy or 6 months after the last dose of paclitaxel. Men participants who are sexually active with women of childbearing potential will be instructed to adhere to contraception and must refrain from sperm donation for a period of 180 days after the last dose of durvalumab and tremelimumab or 90 days after the last dose of durvalumab monotherapy or 6 months after the last dose of paclitaxel.
15. Registration in a national health care system (PUMA included).

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
2. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) or supportive care clinical study or during the follow-up period of an interventional study.
3. Receipt of the last dose of anticancer therapy (investigational product, chemotherapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies) ≤ 21 days prior to the first dose of study drug. If sufficient wash-out time has not occurred due to the schedule or pharmacokinetics properties of an agent, a longer wash-out period will be required, as agreed by AstraZeneca/MedImmune and the investigator.
4. Mixed histology (hepatocholangiocarcinoma).
5. Extensive tumor massively replacing both entire lobes.
6. Obstructive jaundice (bilirubin > 1.5 ULN) without adequate biliary drainage.
7. Any unresolved toxicity NCI CTCAE Grade ≥ 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   * Patients with Grade ≥ 2 neuropathy will be excluded
   * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Physician.
8. History of allogenic organ transplantation.
9. Any systemic steroid therapy (> 10 mg daily dose of prednisone or equivalent) whatever the duration of this corticotherapy

   Note: The following are exceptions to this criterion:
   * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
   * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
   * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
10. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies) Note: Patients with past HBV infection or resolved HBV infection (defined as having a negative HBsAg test and a positive hepatitis B core antigen [HBc] antibody test) are eligible.

    Note: Patients positive for HCV antibody are eligible only if polymerase chain reaction testing is negative for HCV ribonucleic acid (RNA).
11. Diagnosis of any second malignancy within the last 5 years, except for adequately treated basal cell or squamous cell skin cancer, or in situ carcinoma of the cervix uteri.
12. Prior treatment with taxane or any immune ICI, including durvalumab and tremelimumab or any other anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibody.
13. Known active central nervous system metastases and/or carcinomatous meningitis; patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids > 10 mg/day of prednisone or equivalent for at least 14 days prior to trial treatment.
14. Uncontrolled massive pleural effusion or massive ascites.
15. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]), that has required systemic treatment (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs) Note: Patients with vitiligo, alopecia, or any chronic skin condition that does not require systemic therapy are exception to this criterion.

    Note: History of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible.

    Note: Controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible.
16. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
17. Live vaccine administration within 30 days prior to the first dose of study treatment Note: Patients, if enrolled, should not receive live vaccine whilst receiving investigational product and up to 30 days after the last dose of investigational product.
18. Known or suspected allergy or hypersensitivity to any of the study drugs or any of the study drug excipients (taxane, durvalumab, or tremelimumab).
19. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥ 470 ms.
20. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with participation for the full duration of the trial, or is not in the best interest of the participant, in the opinion of the treating investigator.
21. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug.
22. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of investigational product Note: Local surgery of isolated lesions for palliative intent is acceptable.
23. Pregnancy/lactation.
24. Tutelage or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2018-11-09 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) in amended Arm A | At 6 months
  OS - defined as the time from date of randomization to date of death. In the absence of confirmation of death, survival time will be censored at the date of the last clinical assessment

SECONDARY OUTCOMES:
Safety profile - All grade and severe (grade 3-5) | From signature of informed consent to 3 months after last study treatment administration
  All grade and severe (grade 3-5) adevrse events, according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v 5.0
RECIST v1.1 and iRECIST criteria in arm A and amended Arm A | At 2 months, evaluation every 2 months during treatment period and end of treatment (until the date of first documented progression or date of death, assessed up to 30 months
  RECIST v1.1 and iRECIST criteria comparison for tumor response evaluation in arm A and amended Arm A
Health-related Quality of life (HRQoL) assessed by EORTC QLQ-C30 questionnaire in Arm A and amended Arm A | Baseline, every 2 months during treatment period and end of treatment (until the date of first documented progression or date of death)
  A quality of life score is obtained according to the answers to the questionnaires.
Health-related Quality of life (HRQoL) assessed by EORTC QLQ-BIL21 questionnaire | Baseline, every 2 months during treatment period and end of treatment (until the date of first documented progression or date of death)
  A quality of life score is obtained according to the answers to the questionnaires.
Quality-Adjusted Time Without Symptoms of Disease or Toxicity of Treatment (Q-Twist) in arm A and amended Arm A | assessed up to 30 months
  Q-TWiST analysis considers three health states, TOX, TWiST, and REL, and the duration of each state is calculated for every patient.
Predictive markers of response in arm A and amended arm A | Baseline, Month 2, Month 4, Month 8, Month 12, Month 18, Month 24 and end of study (until the date of first documented progression or date of death, assessed up 30 months
  Evaluation of predictive markers of response in arm A and amended arm A
Progression free survival (PFS) in Arm A and Amended Arm A | at 4 months
  PFS at 4 months according to iRECIST (centralized review of CT-scan imaging) Note: disease progression on CT-scan imaging must be confirmed by a new imaging at 4 weeks in order to meet iRECIST criteria.
Overall Survival (OS) in Arm A | At 6 months
  OS - defined as the time from date of randomization to date of death. In the absence of confirmation of death, survival time will be censored at the date of the last clinical assessment

CONTACTS AND LOCATIONS:
Overall Officials: Cindy NEUZILLET, Principal Investigator — Institut Curie site de Saint Cloud
Locations (28):
- France (28):
  - CHRU Jean Minjoz, Besançon
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Hôpital Duchenne, Boulogne-sur-Mer
  - CHU Morvan, Brest
  - Hôpital Beaujon, Clichy
  - CHPSO Site de Creil, Creil
  - CHU Henri Mondor, Créteil
  - Centre Georges François Leclerc, Dijon
  - CHU Dijon, Dijon
  - Institut Andrée Dutreix, Dunkirk
  - Institut Hospitalier franco-Britannique, Levallois-Perret
  - CHRU Lille, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - Hôpital la Timone, Marseille
  - Hôpital Saint Eloi, Montpellier
  - Hôpital Prive du confluent SAS, Nantes
  - Hôpital Cochin, Paris
  - Hôpital Saint Antoine, Paris
  - Institut Mutualiste Montsouris, Paris
  - Hôpital Haut Lévêque, Pessac
  - CHU Poitiers, Poitiers
  - CHU Robert Debré, Reims
  - Centre Eugène Marquis, Rennes
  - Institut Curie, Saint-Cloud
  - CHI Poissy Saint Germain, Saint-Germain-en-Laye
  - Centre Paul Strauss, Strasbourg
  - Insitut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boileve A, Hilmi M, Gougis P, Cohen R, Rousseau B, Blanc JF, Ben Abdelghani M, Castanie H, Dahan L, Tougeron D, Metges JP, Tournigand C, Garcia-Larnicol ML, Vernerey D, Turpin A, Neuzillet C. Triplet combination of durvalumab, tremelimumab, and paclitaxel in biliary tract carcinomas: Safety run-in results of the randomized IMMUNOBIL PRODIGE 57 phase II trial. Eur J Cancer. 2021 Jan;143:55-63. doi: 10.1016/j.ejca.2020.10.027. Epub 2020 Dec 3. PMID 33279854